CLINICAL TRIAL: NCT00432796
Title: A Double Blind Randomized Control Trial of Post-Operative Low Molecular Weight Heparin Bridging Therapy Versus Placebo Bridging Therapy for Patients Who Are at High Risk for Arterial Thromboembolism (PERIOP 2)
Brief Title: PERIOP 2 - A Safety and Effectiveness of LMWH vs Placebo Bridging Therapy for Patients on Long Term Warfarin Requiring Temporary Interruption of Warfarin.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Pfizer (Industry)
Responsible Party: Principal Investigator, Michael Kovacs, M.D., London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R-06-267; NRA6300019
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Stroke
Keywords: Anticoagulation; Prosthetic heart valves; Atrial fibrillation; Bridging Therapy; Thromboembolism; Warfarin; Low Molecular Weight Heparin
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Thromboembolism | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): patients are randomized post-operative to receive either active treatment or placebo.
  Active treatment is Dalteparin injectable. Patients randomized to active treatment will receive Dalteparin 5,000 iu or 200 iu/kg once daily depending on the type of surgery they have had.
  Interventions: Drug: Dalteparin
- 2 (Experimental): patients will be randomized post-operative to receive either active treatment or placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dalteparin — 5,000 iu or 200 iu/kg depending on the type of surgery injection will be given subcutaneously, once a day for a minimum of 4 days or until the INR is 2.0
  Other Names: Fragmin
  Arms: 1
Other: Placebo — patients will be randomized post-operative to receive either active treatment or placebo.
  the placebo will be given as a subcutaneous injection once a day. the amount of the placebo will be equivalent to the active treatment depending on the type of surgery.
  ie. 5,000 iu or 200 iu/kg
  Arms: 2

SUMMARY:
The purpose of the study is to determine the effectiveness and safety of LMWH postoperative bridging therapy (standard of care) versus postoperative placebo bridging therapy (experimental arm)for patients with mechanical heart valves or atrial fibrillation or atrial flutter who are at high risk for stroke when warfarin is temporarily interrupted for a procedure.

DETAILED DESCRIPTION:
There are a growing number of patients who receive long-term warfarin therapy for the prevention of arterial thromboembolism. The current approach to the perioperative management of anticoagulation (i.e. "bridging therapy") with low molecular weight heparin (LMWH) is not standardized and has not been assessed by adequate randomized studies. Most clinicians, however, recommend bridging therapy.

We have recently completed a multicentre single arm pilot study of LMWH bridging therapy. This study in 10 centres accrued 224 patients in 10 months. In the pilot study the postoperative thromboembolic event rate was 3.1% and 75% of these occurred in patients who had anticoagulation held due to bleeding.

Design:A prospective multicentre randomized double-blind controlled trial. Patients: Consecutive eligible and consenting patients from 11 teaching hospitals in Canada. A total of 1773 patients with prosthetic heart valves receiving long-term oral anticoagulation with warfarin or patients with atrial fibrillation/flutter and a major risk factor who require elective non-cardiac surgery or invasive procedure necessitating reversal of their oral anticoagulant therapy.

Treatment Schedule: Consent will be obtained preoperatively but randomization will be performed postoperatively after confirming eligibility.

Preoperative period: In all participants, warfarin therapy will be discontinued five days prior to the procedure. Dalteparin, a LMWH, will be administered at 200 IU/kg sc early in the morning for the three days prior to, but not including the day of, the procedure except on the day prior to surgery the dose will be 100 I.U./kg given 24 hours preoperatively. Warfarin will be resumed the evening of the procedure.

Postoperative period: Dalteparin or placebo will be administered daily (starting the morning after the procedure), provided surgical hemostasis is achieved, and will be continued for at least four days and until the INR is>2.0. Patients considered at high risk for a postoperative major bleed will be given dalteparin or placebo at a dose of 5,000 IU sc daily. Patients who undergo procedures that are considered low risk for bleeding complications will resume dalteparin or placebo at 200 IU/Kg s.c. daily.

Outcomes:The primary outcome will be the frequency of episodes of major thromboembolism over a 90-day follow-up period following the time of randomization. Secondary outcomes will include major bleeding and overall survival.

Relevance: To bridge or not to bridge, is a common clinical question, without randomized trial evidence to guide clinicians. This RCT will answer whether post-operative bridging reduces risk of thromboembolism or causes harm.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent,
2. Patients aged >18
3. Patients with prosthetic(mechanical) heart valve
4. Patients with atrial fibrillation or atrial flutter and a major risk factor (previous TIA or stroke, high blood pressure, diabetes, aged >75, moderate/severe left ventricle dysfunction)
5. Who are receiving long-term oral anticoagulation and require elective non-cardiac surgery or an invasive procedure with reversal of their anticoagulant therapy.

Exclusion Criteria:

1. Evidence of active bleeding within last 30 days prior to stopping warfarin.
2. Platelet count <100 x 109/L.
3. Spinal or neurosurgery.
4. Life expectancy less than 3 months.
5. Calculated creatinine clearance <30 ml/min
6. Patients requiring cardiac surgery.
7. Multiple prosthetic(mechanical) valves or Starr-Edwards valve or prosthetic(mechanical) valve with a history of stroke or TIA
8. History of heparin induced thrombocytopenia (HIT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1473 (Actual)
Dates: Start 2006-12; Primary Completion 2019-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
major thromboembolism | 90 days from randomization

SECONDARY OUTCOMES:
major bleeding | 90 days from randomization
minor bleeding | 90 days from randomization
a composite of major bleeding and major thromboembolic events | 90 days from randomization
minor thromboembolic events | 90 days from randomization
overall survival. | 90 days from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Kovacs, MD, FRCPC, Principal Investigator — University of Western Ontario, Canada
Locations (8):
- Canada (6):
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation-General Hospital, Hamilton, Ontario
  - Hamilton Health Sciences Corporation-McMaster Site, Hamilton, Ontario
  - Hamilton Health Sciences Corporation-Henderson Site, Hamilton, Ontario
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec
- India (2):
  - Care Hospital, Hyderabad, Nampally
  - Sir Ganga Ram Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tu JV, Gong Y. Trends in treatment and outcomes for acute stroke patients in Ontario, 1992-1998. Arch Intern Med. 2003 Feb 10;163(3):293-7. doi: 10.1001/archinte.163.3.293. PMID 12578509
- [Background] Kearon C, Hirsh J. Management of anticoagulation before and after elective surgery. N Engl J Med. 1997 May 22;336(21):1506-11. doi: 10.1056/NEJM199705223362107. No abstract available. PMID 9154771
- [Background] Vongpatanasin W, Hillis LD, Lange RA. Prosthetic heart valves. N Engl J Med. 1996 Aug 8;335(6):407-16. doi: 10.1056/NEJM199608083350607. No abstract available. PMID 8676934
- [Background] Cannegieter SC, Rosendaal FR, Briet E. Thromboembolic and bleeding complications in patients with mechanical heart valve prostheses. Circulation. 1994 Feb;89(2):635-41. doi: 10.1161/01.cir.89.2.635. PMID 8313552
- [Background] White RH, McKittrick T, Hutchinson R, Twitchell J. Temporary discontinuation of warfarin therapy: changes in the international normalized ratio. Ann Intern Med. 1995 Jan 1;122(1):40-2. doi: 10.7326/0003-4819-122-1-199501010-00006. PMID 7985894
- [Background] Kovacs MJ, Rodger M, Anderson DR, Morrow B, Kells G, Kovacs J, Boyle E, Wells PS. Comparison of 10-mg and 5-mg warfarin initiation nomograms together with low-molecular-weight heparin for outpatient treatment of acute venous thromboembolism. A randomized, double-blind, controlled trial. Ann Intern Med. 2003 May 6;138(9):714-9. doi: 10.7326/0003-4819-138-9-200305060-00007. PMID 12729425
- [Background] Madura JA, Rookstool M, Wease G. The management of patients on chronic Coumadin therapy undergoing subsequent surgical procedures. Am Surg. 1994 Jul;60(7):542-6; discussion 546-7. PMID 8010570
- [Background] Eckman MH, Beshansky JR, Durand-Zaleski I, Levine HJ, Pauker SG. Anticoagulation for noncardiac procedures in patients with prosthetic heart valves. Does low risk mean high cost? JAMA. 1990 Mar 16;263(11):1513-21. PMID 2106590
- [Background] Katholi RE, Nolan SP, McGuire LB. The management of anticoagulation during noncardiac operations in patients with prosthetic heart valves. A prospective study. Am Heart J. 1978 Aug;96(2):163-5. doi: 10.1016/0002-8703(78)90080-7. PMID 676976
- [Background] Stein PD, Alpert JS, Copeland J, Dalen JE, Goldman S, Turpie AG. Antithrombotic therapy in patients with mechanical and biological prosthetic heart valves. Chest. 1995 Oct;108(4 Suppl):371S-379S. doi: 10.1378/chest.108.4_supplement.371s. No abstract available. PMID 7555190
- [Background] Douketis JD, Crowther MA, Cherian SS, Kearon CB. Physician preferences for perioperative anticoagulation in patients with a mechanical heart valve who are undergoing elective noncardiac surgery. Chest. 1999 Nov;116(5):1240-6. doi: 10.1378/chest.116.5.1240. PMID 10559081
- [Background] Dunn AS, Turpie AG. Perioperative management of patients receiving oral anticoagulants: a systematic review. Arch Intern Med. 2003 Apr 28;163(8):901-8. doi: 10.1001/archinte.163.8.901. PMID 12719198
- [Background] Douketis JD, Johnson JA, Turpie AG. Low-molecular-weight heparin as bridging anticoagulation during interruption of warfarin: assessment of a standardized periprocedural anticoagulation regimen. Arch Intern Med. 2004 Jun 28;164(12):1319-26. doi: 10.1001/archinte.164.12.1319. PMID 15226166
- [Background] Spandorfer JM, Lynch S, Weitz HH, Fertel S, Merli GJ. Use of enoxaparin for the chronically anticoagulated patient before and after procedures. Am J Cardiol. 1999 Aug 15;84(4):478-80, A10. doi: 10.1016/s0002-9149(99)00341-0. PMID 10468095
- [Background] Kovacs MJ, Kearon C, Rodger M, Anderson DR, Turpie AG, Bates SM, Desjardins L, Douketis J, Kahn SR, Solymoss S, Wells PS. Single-arm study of bridging therapy with low-molecular-weight heparin for patients at risk of arterial embolism who require temporary interruption of warfarin. Circulation. 2004 Sep 21;110(12):1658-63. doi: 10.1161/01.CIR.0000142859.77578.C9. Epub 2004 Sep 13. PMID 15364803
- [Background] Ferreira I, Dos L, Tornos P, Nicolau I, Permanyer-Miralda G, Soler-Soler J. Experience with enoxaparin in patients with mechanical heart valves who must withhold acenocumarol. Heart. 2003 May;89(5):527-30. doi: 10.1136/heart.89.5.527. PMID 12695457
- [Background] Omran H, Hammerstingl C, Schmidt H, von der Recke G, Paar WD, Luderitz B. A prospective and randomized comparison of the safety and effects of therapeutic levels of enoxaparin versus unfractionated heparin in chronically anticoagulated patients undergoing elective cardiac catheterization. Thromb Haemost. 2003 Aug;90(2):267-71. doi: 10.1160/TH02-10-0159. PMID 12888874
- [Background] Tinmouth AH, Morrow BH, Cruickshank MK, Moore PM, Kovacs MJ. Dalteparin as periprocedure anticoagulation for patients on warfarin and at high risk of thrombosis. Ann Pharmacother. 2001 Jun;35(6):669-74. doi: 10.1345/aph.10305. PMID 11408982
- [Background] POLLER L, THOMSON J. EVIDENCE FOR
- [Background] Grip L, Blomback M, Schulman S. Hypercoagulable state and thromboembolism following warfarin withdrawal in post-myocardial-infarction patients. Eur Heart J. 1991 Nov;12(11):1225-33. doi: 10.1093/eurheartj/12.11.1225. PMID 1782954
- [Background] Palareti G, Legnani C, Guazzaloca G, Frascaro M, Grauso F, De Rosa F, Fortunato G, Coccheri S. Activation of blood coagulation after abrupt or stepwise withdrawal of oral anticoagulants--a prospective study. Thromb Haemost. 1994 Aug;72(2):222-6. PMID 7831656
- [Background] Valles J, Aznar J, Santos T, Villa P, Fernandez A. Platelet function in patients with chronic coronary heart disease on long-term anticoagulant therapy: effect of anticoagulant stopping. Haemostasis. 1993 Jul-Aug;23(4):212-8. doi: 10.1159/000216877. PMID 8314171
- [Background] Raskob GE, Durica SS, Morrissey JH, Owen WL, Comp PC. Effect of treatment with low-dose warfarin-aspirin on activated factor VII. Blood. 1995 Jun 1;85(11):3034-9. PMID 7756639
- [Background] Genewein U, Haeberli A, Straub PW, Beer JH. Rebound after cessation of oral anticoagulant therapy: the biochemical evidence. Br J Haematol. 1996 Feb;92(2):479-85. doi: 10.1046/j.1365-2141.1996.d01-1499.x. PMID 8603020
- [Background] Adjusted-dose warfarin versus low-intensity, fixed-dose warfarin plus aspirin for high-risk patients with atrial fibrillation: Stroke Prevention in Atrial Fibrillation III randomised clinical trial. Lancet. 1996 Sep 7;348(9028):633-8. PMID 8782752
- [Background] Weitz JI. Low-molecular-weight heparins. N Engl J Med. 1997 Sep 4;337(10):688-98. doi: 10.1056/NEJM199709043371007. No abstract available. PMID 9278467
- [Background] Kovacs MJ, Weir K, MacKinnon K, Keeney M, Brien WF, Cruickshank MK. Body weight does not predict for anti-Xa levels after fixed dose prophylaxis with enoxaparin after orthopedic surgery. Thromb Res. 1998 Aug 1;91(3):137-42. doi: 10.1016/s0049-3848(98)00083-8. PMID 9733157
- [Background] Cohen M, Demers C, Gurfinkel EP, Turpie AG, Fromell GJ, Goodman S, Langer A, Califf RM, Fox KA, Premmereur J, Bigonzi F. A comparison of low-molecular-weight heparin with unfractionated heparin for unstable coronary artery disease. Efficacy and Safety of Subcutaneous Enoxaparin in Non-Q-Wave Coronary Events Study Group. N Engl J Med. 1997 Aug 14;337(7):447-52. doi: 10.1056/NEJM199708143370702. PMID 9250846
- [Background] Low-molecular-weight heparin during instability in coronary artery disease, Fragmin during Instability in Coronary Artery Disease (FRISC) study group. Lancet. 1996 Mar 2;347(9001):561-8. PMID 8596317
- [Background] Levine M, Gent M, Hirsh J, Leclerc J, Anderson D, Weitz J, Ginsberg J, Turpie AG, Demers C, Kovacs M. A comparison of low-molecular-weight heparin administered primarily at home with unfractionated heparin administered in the hospital for proximal deep-vein thrombosis. N Engl J Med. 1996 Mar 14;334(11):677-81. doi: 10.1056/NEJM199603143341101. PMID 8594425
- [Background] Koopman MM, Prandoni P, Piovella F, Ockelford PA, Brandjes DP, van der Meer J, Gallus AS, Simonneau G, Chesterman CH, Prins MH. Treatment of venous thrombosis with intravenous unfractionated heparin administered in the hospital as compared with subcutaneous low-molecular-weight heparin administered at home. The Tasman Study Group. N Engl J Med. 1996 Mar 14;334(11):682-7. doi: 10.1056/NEJM199603143341102. PMID 8594426
- [Background] Columbus Investigators; Buller HR, Gent M, Gallus AS, Ginsberg J, Prins MH, Baildon R. Low-molecular-weight heparin in the treatment of patients with venous thromboembolism. N Engl J Med. 1997 Sep 4;337(10):657-62. doi: 10.1056/NEJM199709043371001. PMID 9280815
- [Background] Simonneau G, Sors H, Charbonnier B, Page Y, Laaban JP, Azarian R, Laurent M, Hirsch JL, Ferrari E, Bosson JL, Mottier D, Beau B. A comparison of low-molecular-weight heparin with unfractionated heparin for acute pulmonary embolism. The THESEE Study Group. Tinzaparine ou Heparine Standard: Evaluations dans l'Embolie Pulmonaire. N Engl J Med. 1997 Sep 4;337(10):663-9. doi: 10.1056/NEJM199709043371002. PMID 9278462
- [Background] Schafer AI, Levine MN, Konkle BA, Kearon C. Thrombotic disorders: diagnosis and treatment. Hematology Am Soc Hematol Educ Program. 2003:520-39. doi: 10.1182/asheducation-2003.1.520. PMID 14633797
- [Background] Hirsh J, Raschke R. Heparin and low-molecular-weight heparin: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):188S-203S. doi: 10.1378/chest.126.3_suppl.188S. PMID 15383472
- [Background] Geerts WH, Pineo GF, Heit JA, Bergqvist D, Lassen MR, Colwell CW, Ray JG. Prevention of venous thromboembolism: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):338S-400S. doi: 10.1378/chest.126.3_suppl.338S. PMID 15383478
- [Background] Kearon C, Hirsh J. Perioperative management of patients receiving oral anticoagulants. Arch Intern Med. 2003 Nov 10;163(20):2532-3; author reply 2533. doi: 10.1001/archinte.163.20.2532-b. No abstract available. PMID 14609792
- [Background] Risk factors for stroke and efficacy of antithrombotic therapy in atrial fibrillation. Analysis of pooled data from five randomized controlled trials. Arch Intern Med. 1994 Jul 11;154(13):1449-57. PMID 8018000
- [Background] Crowther MA, Julian J, McCarty D, Douketis J, Kovacs M, Biagoni L, Schnurr T, McGinnis J, Gent M, Hirsh J, Ginsberg J. Treatment of warfarin-associated coagulopathy with oral vitamin K: a randomised controlled trial. Lancet. 2000 Nov 4;356(9241):1551-3. doi: 10.1016/S0140-6736(00)03125-1. PMID 11075768
- [Background] Kearon C, Ginsberg JS, Kovacs MJ, Anderson DR, Wells P, Julian JA, MacKinnon B, Weitz JI, Crowther MA, Dolan S, Turpie AG, Geerts W, Solymoss S, van Nguyen P, Demers C, Kahn SR, Kassis J, Rodger M, Hambleton J, Gent M; Extended Low-Intensity Anticoagulation for Thrombo-Embolism Investigators. Comparison of low-intensity warfarin therapy with conventional-intensity warfarin therapy for long-term prevention of recurrent venous thromboembolism. N Engl J Med. 2003 Aug 14;349(7):631-9. doi: 10.1056/NEJMoa035422. PMID 12917299
- [Background] Crowther MA, Ginsberg JS, Julian J, Denburg J, Hirsh J, Douketis J, Laskin C, Fortin P, Anderson D, Kearon C, Clarke A, Geerts W, Forgie M, Green D, Costantini L, Yacura W, Wilson S, Gent M, Kovacs MJ. A comparison of two intensities of warfarin for the prevention of recurrent thrombosis in patients with the antiphospholipid antibody syndrome. N Engl J Med. 2003 Sep 18;349(12):1133-8. doi: 10.1056/NEJMoa035241. PMID 13679527
- [Background] Wilson JT, Hareendran A, Grant M, Baird T, Schulz UG, Muir KW, Bone I. Improving the assessment of outcomes in stroke: use of a structured interview to assign grades on the modified Rankin Scale. Stroke. 2002 Sep;33(9):2243-6. doi: 10.1161/01.str.0000027437.22450.bd. PMID 12215594
- [Background] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593
- [Background] Rodger M, Bredeson C, Wells PS, Beck J, Kearns B, Huebsch LB. Cost-effectiveness of low-molecular-weight heparin and unfractionated heparin in treatment of deep vein thrombosis. CMAJ. 1998 Oct 20;159(8):931-8. PMID 9834718
- [Background] Buller HR, Davidson BL, Decousus H, Gallus A, Gent M, Piovella F, Prins MH, Raskob G, van den Berg-Segers AE, Cariou R, Leeuwenkamp O, Lensing AW; Matisse Investigators. Subcutaneous fondaparinux versus intravenous unfractionated heparin in the initial treatment of pulmonary embolism. N Engl J Med. 2003 Oct 30;349(18):1695-702. doi: 10.1056/NEJMoa035451. PMID 14585937
- [Derived] Kovacs MJ, Wells PS, Anderson DR, Lazo-Langner A, Kearon C, Bates SM, Blostein M, Kahn SR, Schulman S, Sabri E, Solymoss S, Ramsay T, Yeo E, Rodger MA; PERIOP2 Investigators. Postoperative low molecular weight heparin bridging treatment for patients at high risk of arterial thromboembolism (PERIOP2): double blind randomised controlled trial. BMJ. 2021 Jun 9;373:n1205. doi: 10.1136/bmj.n1205. PMID 34108229